CLINICAL TRIAL: NCT04551326
Title: Immediate Effect of Hamstring Stretching in Patients With Chronic Low Back Pain
Acronym: EFIM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 DOBIJA; 2019-A03000-57 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-02

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic low back pain; Hamstring flexibility; Hamstring stretching; Immediate stretching effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hamstring stretching (Experimental): Participants' lower limb will be positioned in maximal hip flexion and gradually moved to maximal knee extension by physical therapist. The procedure will take one minute for each lower limb.
  Interventions: Other: manual hamstring stretching

INTERVENTIONS:
Other: manual hamstring stretching — Participants' lower limb will be positioned in maximal hip flexion and gradually moved to maximal knee extension by physical therapist. The procedure will take one minute for each lower limb.

SUMMARY:
Thigh muscles flexibility deficits contribute to handicap in chronic low back pain patients. The study aims to evaluate the immediate effect of thigh muscles stretching in patients with chronic low back pain. The investigation team suppose that flexibility improvement could be detected by instrumented clinical measurements and such difference could be related to psycho-social factors evaluated by questionnaires.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the immediate effect of the hamstring muscle stretching in patients presenting chronic low back pain. The secondary objectives are: (1) to evaluate intra- and interrater reliability, construct validity and responsiveness of the hamstring flexibility measurements (Active Knee Extension [AKE], Straight Leg Rise [SLR]) realised with digital inclinometer, (2) to evaluate factors that potentially could influence immediate effect of the hamstring stretching, specifically psycho-social factors Fear Avoidance Belief Questionnaire (FABQ), Hospital Anxiety and Depression scale (HAD), neuropathic pain presence (DN4).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Chronic low back pain (>3 months) with or without pain irradiation to lower limb
* Hamstring flexibility deficit (AKE <80° and FTF>5cm)

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Condition of restricted mental/legal autonomy (ex. guardianship) ,
* No social security insurance,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension test (AKE) | Day 1
  Description: Participant positioned in supine lying will actively extend his knee while keeping his hip joint in 90 degrees of flexion. Hip position will be verified by digital inclinometer and maintained with a barre indicating vertical position of the participants' thigh. The range of motion will be recorded with digital inclinometer positioned on the tibial craft of the exanimated limb.

SECONDARY OUTCOMES:
Straight Leg Rise test (SLR) | Day 1 before stretching, Day 1 after stretching
  Participant positioned in supine lying, examiner rise his lower limb, with knee extended. Examiner stops the movement when participant declare pain or tension onset than the range of motion is recorded in degree with digital inclinometer positioned on the tibial craft of the exanimated limb.
Fingertip-to-floor distance (FTF) | Day 1 before stretching, Day 1 after stretching
  Participant try to reach the floor with his fingertip by bending forward in the same time knees are kept extended. The distance between fingertips and floor are measured in centimetres by examiner.
Fear Avoidance Belief Questionnaire (FABQ) | Day 1
  Questionnaire evaluating belief about physical activity and work activity. The The FABQ is divided into 2 parts, (1)physical activity (minimum score 0, maximum score 24) and (2) work (minimum score 0, maximum score 42). A higher score indicates more strongly held fear avoidance beliefs.
Ostwestry Disability Index | Day 1
  Questionnaire evaluating pain and function in low back pain patients. Maximum score 100%, minimum score 0%, A higher score indicates greater disability.
Anxiety and Depression scale | Day 1
  Questionnaire evaluating anxiety and depression, Hospital Anxiety and Depression scale. The scale is devided into 2 parts: (1) anxiety (minimum score 0, maximum sore 21) and (2) depression (minimum score 0, maximum sore 21). A higher score indicates greater anxiety or greater depression.
Neuropathic pain presence | Day 1
  Questionnaire evaluating existence of the neuropathic pain, Neuropathic pain presence (DN4). Minimum score 0, maximum sore 10. The score equal or superior to 4 indicate the presence of neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital, Clermont Ferrand, Clermont-Ferrand
  - CHu de Nîmes, Nîmes